CLINICAL TRIAL: NCT00773123
Title: Efficacy of Retinal Nerve Fiber Layer (RNFL) / Ganglion Cell Layer Thickness Ratio by RT-View Utilizing Spectral -Domain Technology as a Diagnostic Predictor of Glaucoma.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Kim,Chan Yun, Institute of Vision Research, Department of Ophthalmology, Severance Hospital, Yonsei University School of Medicine
Other Study IDs: 08-0342
Record Dates: First submitted 2008-10-15; First posted 2008-10-16 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Primary Open Angle Glaucoma
Keywords: RT-View; Spectral domain OCT; Ganglion cell layer; RNFL; Visual field defect
MeSH Terms: conditions — Glaucoma, Open-Angle

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: Primary open angle glaucoma
- 2: Normal controls

SUMMARY:
RT-View utilizes spectral domain technology to assess both RNFL and ganglion cell layer thickness. This study aims to correlate visual field defects in patients with glaucoma to both RNFL and ganglion cell layer thickness.

ELIGIBILITY:
Exclusion Criteria:

* Evidence of retinal disease
* Neovascular glaucoma
* Secondary glaucoma due to intraocular inflammation
* Lens induced glaucoma
* Tumor induced glaucoma

Ages: 10 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: primary open angle glaucoma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-10; Primary Completion 2008-12 (Estimated); Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Ganglion cell layer thickness | 1 month

SECONDARY OUTCOMES:
Visual field defect | 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Vision Research, Department of Ophthalmology, Severance Hospital, Yonsei University School of Medicine, Seoul, South Korea